CLINICAL TRIAL: NCT03060603
Title: Proliferative Effects of Erythropoietin on Human Endometrium
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Collaborators: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, MEHMET AKIF SARGIN, Principal Investigator, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSM EAH-KAEK 2016/7
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Anemia; Endometrial Diseases
Keywords: Erythropoietin; Endometrium; Doppler Ultrasonography
MeSH Terms: conditions — Anemia; Uterine Diseases | interventions — Erythropoietin; Epoetin Alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Erythropoietin: Recombinant Human Erythropoietin, EPREX 4000 IU/0.4 ml, three times in a week, until the correction of anemia, approximately two months.
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — Recombinant Human Erythropoietin, three times in a week, until the correction of anemia, approximately two months.
  Other Names: Recombinant Human Erythropoietin, EPREX 4000 IU/0.4 ml

SUMMARY:
The purpose of this study to assess the proliferative effects of erythropoetin on human endometrium tissue by measuring the endometrial thickness, uterine artery and subendometrial blood flow in postmenopausal women.

DETAILED DESCRIPTION:
20 postmenopausal women who are planned to treat with erythropoietin alpha for their renal conditions will be included to the study. Sample size was calculated with proper power analysis with accepting the difference of 1 mm in endometrial thickness as a significant change. After the informed consent, endometrial thickness (mm), uterine artery and subendometrial blood flow by doppler ultrasonography (RI, S/D) will be measured. Same measurements will be repeated on the 3rd day and 30th day. Patients' age, BMI, co-morbidities, administered erythropoietin doses will be noted. No adverse effect is expected with regard to the ultrasonographic examination. Date of the patients who do not attend for the appointments for repetitive examinations and uninterpretable doppler variables due to the atrophic uterus will be noted as the missing data and will be excluded from the study. Proper statistical analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

* Clinically condition with need for erythropoietin treatment such as anemia due to the renal failure or the need for hemodialysis.
* Must be in postmenopausal period

Exclusion Criteria:

* Patients with any type of malignancy
* Existence of any intracavitary mass which may affect endometrial thickness or blood flow such as endometrial polyps, myomas, intracavitary fluid etc.
* Intrauterine device
* Being on Hormon replacement therapy
* Hysterectomized patients

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients will be recruited from a tertiary research clinic, department of nephrology, Istanbul, Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Endometrial Thickness Confirmed by Transvaginal Ultrasonography at 3th and 30th Days | within the first 3 and 30 days (plus or minus 3 days) after the erythropoietin treatment
  Change from Baseline Endometrial Thickness Confirmed by Transvaginal

CONTACTS AND LOCATIONS:
Overall Officials: Niyazi Tug, Ass.Prof., Study Chair — Executive and Educational Supervisor
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tug N, Altunkaynak ME, Aktas RG, Kilic U, Yilmaz B, Cam C, Karateke A. Does erythropoietin affect motility of spermatozoa? Arch Gynecol Obstet. 2010 May;281(5):933-8. doi: 10.1007/s00404-009-1289-4. Epub 2009 Nov 25. PMID 19937447
- [Background] Tug N, Kilic U, Karateke A, Yilmaz B, Ugur M, Kilic E. Erythropoietin receptor-like immunostaining on human spermatozoa. Reprod Biomed Online. 2010 Nov;21(5):718-20. doi: 10.1016/j.rbmo.2010.05.022. Epub 2010 Jun 19. PMID 20884294
- [Background] Wang L, Di L, Noguchi CT. Erythropoietin, a novel versatile player regulating energy metabolism beyond the erythroid system. Int J Biol Sci. 2014 Aug 23;10(8):921-39. doi: 10.7150/ijbs.9518. eCollection 2014. PMID 25170305
- [Background] Ogilvie M, Yu X, Nicolas-Metral V, Pulido SM, Liu C, Ruegg UT, Noguchi CT. Erythropoietin stimulates proliferation and interferes with differentiation of myoblasts. J Biol Chem. 2000 Dec 15;275(50):39754-61. doi: 10.1074/jbc.M004999200. PMID 10995753
- [Background] Yokomizo R, Matsuzaki S, Uehara S, Murakami T, Yaegashi N, Okamura K. Erythropoietin and erythropoietin receptor expression in human endometrium throughout the menstrual cycle. Mol Hum Reprod. 2002 May;8(5):441-6. doi: 10.1093/molehr/8.5.441. PMID 11994541
- [Result] Yasuda Y, Masuda S, Chikuma M, Inoue K, Nagao M, Sasaki R. Estrogen-dependent production of erythropoietin in uterus and its implication in uterine angiogenesis. J Biol Chem. 1998 Sep 25;273(39):25381-7. doi: 10.1074/jbc.273.39.25381. PMID 9738005